CLINICAL TRIAL: NCT01848015
Title: Prediction of Recurrence in Advanced Gastric Cancer After Radical Resection by Circulating Tumor Cells （CTCs）
Brief Title: Circulating Tumor Cells (CTCs) in Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Other Study IDs: CGOG5003
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
Keywords: CTCs before and after gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- CTCs positive
  Interventions: Other: detection of CTCs

INTERVENTIONS:
Other: detection of CTCs

SUMMARY:
To assess the predictive value of circulating tumor cells (CTCs) for recurrence of advanced gastric cancer after radical resection.

To identify the relationship between the detection of circulation tumor cells and recurrence patterns of gastric cancer after radical resection.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* Preoperative clinical examination and imaging indicating operable disease
* complete resection (R0 resection)
* D2 or D2+ resection

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Patients who have been given preoperative chemotherapy/chemoradiation.
* Staging investigations or intraoperative exploration indicating inoperable disease
* R1 or R2 resection
* D0 or D1 resection
* Patients unreliable for follow up
* Past history of malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with advanced gastric cancer accepted radical resection(D2)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
CTCs | 2 months

SECONDARY OUTCOMES:
Recurrence of gastric cancer after radical resection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, PhD, Principal Investigator — Peking University
Locations (1):
- Peking cancer hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Q, Shan F, Li Z, Gao J, Li Y, Shen L, Ji J, Lu M. A prospective study on the changes and clinical significance of pre-operative and post-operative circulating tumor cells in resectable gastric cancer. J Transl Med. 2018 Jun 20;16(1):171. doi: 10.1186/s12967-018-1544-1. PMID 29925382